CLINICAL TRIAL: NCT06321406
Title: Effect of Superficial Neuromuscular Stimulation on Ultrasonographic Findings of Oropharyngeal Swallowing in Post-stroke Dysphagic Patients.
Brief Title: Effect of Superficial Neuromuscular Stimulation in Post-stroke Dysphagic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Çalış, Professor Doctor, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KayseriCHdysphagia
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Dysphagia; Stroke
Keywords: dysphagia; post-stroke dysphagia; rehabilitation; ultrasonography
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Exercises such as progressively resistant oral-facial, lingual, laryngeal exercises, tongue strengthening exercises, effortful swallowing maneuver, thermal/tactile stimulation to oropharyngeal muscles, Masako maneuver, Mendelson maneuver, Shaker maneuver, which are included in traditional swallowing treatment, will be taught and practiced for 30 minutes will be recommended for one month.
  Interventions: Behavioral: Exercise
- NMES(neuromuscular electrical stimulation) Group (Active Comparator): One electrode will be connected to the suprahyoid region and the other electrode will be connected between the thyroid and hyoid cartilages. Superficial neuromuscular stimulation will be applied by the physiotherapist at 80 Hz, 0-25 µA current range for 20 minutes, for 5 days for the patient, for a total of 4 weeks. At the same time, each patient will be taught the exercises included in traditional swallowing treatment and will be advised to practice them for 30 minutes every day.
  Interventions: Device: NMES (neuromuscular electrical stimulation); Behavioral: Exercise

INTERVENTIONS:
Device: NMES (neuromuscular electrical stimulation) — With this application, swallowing muscles are stimulated and muscle strength increases.
  Arms: NMES(neuromuscular electrical stimulation) Group
Behavioral: Exercise — Traditional Conservative swallowing treatment

SUMMARY:
Swallowing disorder in stroke patients is a significant cause of morbidity and mortality as it can cause aspiration pneumonia. Electrical stimulation has proven to be effective in post-stroke dysphagic patients.10 patients who have symptoms of post-stroke dysphagia, meet the inclusion criteria and volunteer to participate will be included in the study. Included patients will be randomized into 2 groups. The exercise program will be applied to both groups as a home program for 4 weeks.

DETAILED DESCRIPTION:
A randomized, prospective, controlled study will include 10 patients with post-stroke dysphagia. Groups will be randomized into 2 groups.

1. st group; One electrode will be connected to the suprahyoid region and the other electrode will be connected between the thyroid and hyoid cartilages. Superficial neuromuscular stimulation will be applied by the physiotherapist at 80 Hz, 0-25 µA (microampere) current range for 20 minutes, for 5 days for the patient, for a total of 4 weeks. At the same time, each patient will be taught the exercises included in traditional swallowing treatment and will be advised to practice them for 30 minutes every day.
2. nd group; Exercises such as progressively resistant oral-facial, lingual, laryngeal exercises, tongue strengthening exercises, effortful swallowing maneuver, thermal/tactile stimulation to oropharyngeal muscles, Masako maneuver, Mendelson maneuver, Shaker maneuver, which are included in traditional swallowing treatment, will be taught and practiced for 30 minutes will be recommended for one month.

Patients' dysphagia scales, quality of life survey and ultrasonography measurements will be performed before and after treatment.

Tests to be applied

* Functional Oral Intake Scale (FOAS)
* Swallowing Function Screening Test (EAT-10)
* GUSS (Gagging Swallowing Screening Test)
* Modified Mann Swallowing Ability Assessment Test (MMASA)
* SWAL-QOL (The impact of swallowing disorders on quality of life questionnaire),
* Measurements made by ultrasonography (measurement of tongue thickness, measurement of hyoid-larynx distance and measurements of other anatomical structures)

Clinic Responsible for Research: Physical Therapy and Rehabilitation Clinic of Kayseri City Hospital

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over 40 years of age with post-stroke dysphagia
* Patients with Functional Oral Intake Scale (FOAS) 1-6

Exclusion Criteria:

* Patients younger than 40 years old
* Dementia, impaired consciousness or hypoesthetic /anesthetic patients
* Patients with low body mass
* Patients with pacemakers and severe heart disease
* Severe hypertension and hypotension
* Thrombosis or thrombophlebitis
* Pregnancy
* Epilepsy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic measurements | at baseline, 4th week
  Measurements made by ultrasonography (measurement of tongue thickness, measurement of hyoid-larynx distance and measurements of other anatomical structures)

SECONDARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | at baseline, 4th week
  Functional Oral Intake Scale (FOIS) is an ordinal scale with validity and reliability designed to evaluate the current status and functional change in oral intake of patients with neurogenic dysphagia. This scale consists of 7 items. Items 1 to 3 are related to inability to feed orally, items 4 to 7 are related to oral feeding.
Swallowing Function Screening Test (EAT-10) | at baseline, 4th week
  It is a useful questionnaire consisting of 10 questions with Turkish validity and reliability and which patients can easily fill out.
GUSS (Gagging Swallowing Screening Test) | at baseline, 4th week
  GUSS is one of the approved swallowing screening tests in acute stroke patients. It provides dietary recommendations as well as screening for aspiration risk. It consists of two main parts; In the first part, conditions such as alertness, salivation, and cough are evaluated as an indirect swallowing test. In the second part, the direct swallowing test, swallowing trials are performed with three different consistencies: semi-solid, liquid and solid. 5 points are achieved in each subgroup. Scores between 0 and 9 are considered as severe dysphagia and special diet and videofluoroscopic examination are recommended. 10-14 points are considered moderate dysphagia, 5-19 points are considered mild dysphagia, and 20 points are considered normal.
Modified Mann Swallowing Ability Assessment Test (MMASA) | at baseline, 4th week
  It is a bedside test that evaluates parameters such as alertness, cooperation, respiration, expressive speech, auditory perception, dysarthria, salivation, tongue movement, tongue strength, gagging, cough reflex and palate movement. The highest score is 100. It is recommended that patients who score 94 or below as a result of the evaluation should not be fed orally and should be referred to a speech-language pathologist.
SWAL-QOL (The impact of swallowing disorders on quality of life questionnaire) | at baseline, 4th week
  Swallow Quality of Life Questionnaire (SWAL-QOL) is one of the most widely known patient based and dysphagia specific item questionnaire. It is a valid and reliable scale in the evaluation of dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan YAĞMUR GÖZ, Principal Investigator — Kayseri City Hospital
Locations (1):
- health sciences university Kayseri medicine faculty, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Cook IJ, Kahrilas PJ. AGA technical review on management of oropharyngeal dysphagia. Gastroenterology. 1999 Feb;116(2):455-78. doi: 10.1016/s0016-5085(99)70144-7. No abstract available. PMID 9922328
- [Background] Kuhl V, Eicke BM, Dieterich M, Urban PP. Sonographic analysis of laryngeal elevation during swallowing. J Neurol. 2003 Mar;250(3):333-7. doi: 10.1007/s00415-003-1007-2. PMID 12638025
- [Background] Bath PM, Lee HS, Everton LF. Swallowing therapy for dysphagia in acute and subacute stroke. Cochrane Database Syst Rev. 2018 Oct 30;10(10):CD000323. doi: 10.1002/14651858.CD000323.pub3. PMID 30376602
- [Background] Simonelli M, Ruoppolo G, Iosa M, Morone G, Fusco A, Grasso MG, Gallo A, Paolucci S. A stimulus for eating. The use of neuromuscular transcutaneous electrical stimulation in patients affected by severe dysphagia after subacute stroke: A pilot randomized controlled trial. NeuroRehabilitation. 2019;44(1):103-110. doi: 10.3233/NRE-182526. PMID 30714980
- [Background] Chiang CF, Lin MT, Hsiao MY, Yeh YC, Liang YC, Wang TG. Comparative Efficacy of Noninvasive Neurostimulation Therapies for Acute and Subacute Poststroke Dysphagia: A Systematic Review and Network Meta-analysis. Arch Phys Med Rehabil. 2019 Apr;100(4):739-750.e4. doi: 10.1016/j.apmr.2018.09.117. Epub 2018 Oct 21. PMID 30352222
- [Background] Konecny P, Elfmark M. Electrical stimulation of hyoid muscles in post-stroke dysphagia. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2018 Mar;162(1):40-42. doi: 10.5507/bp.2017.043. Epub 2017 Nov 2. PMID 29097820
- [Background] Lim KB, Lee HJ, Lim SS, Choi YI. Neuromuscular electrical and thermal-tactile stimulation for dysphagia caused by stroke: a randomized controlled trial. J Rehabil Med. 2009 Feb;41(3):174-8. doi: 10.2340/16501977-0317. PMID 19229451
- [Background] Oh DH, Park JS, Kim HJ, Chang MY, Hwang NK. The effect of neuromuscular electrical stimulation with different electrode positions on swallowing in stroke patients with oropharyngeal dysphagia: A randomized trial. J Back Musculoskelet Rehabil. 2020;33(4):637-644. doi: 10.3233/BMR-181133. PMID 31594198
- [Background] Robbins J, Kays SA, Gangnon RE, Hind JA, Hewitt AL, Gentry LR, Taylor AJ. The effects of lingual exercise in stroke patients with dysphagia. Arch Phys Med Rehabil. 2007 Feb;88(2):150-8. doi: 10.1016/j.apmr.2006.11.002. PMID 17270511